CLINICAL TRIAL: NCT01289561
Title: Combined Effects of Alcohol and Caffeine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland Griffiths, Professor, Department of Psychiatry,, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00036826; 5R01DA003890-25 (NIH)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Alcohol or Other Drugs Effects
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alcohol self-administration (Experimental): All participants will participate in seven sessions. In three sessions, each participant will consume a beverage containing alcohol and caffeine. In three separate sessions, participants will consume a beverage containing alcohol and caffeine-placebo. In the final session, all participants may choose which beverage they consume. Participants and research assistants will be blinded to inclusion of caffeine/caffeine-placebo in beverage, but each beverage will be labeled for identification (e.g., A or B).
  Interventions: Drug: Alcohol + Caffeine Beverage; Drug: Alcohol + Caffeine-placebo

INTERVENTIONS:
Drug: Alcohol + Caffeine Beverage — 14 g alcohol per 180 ml total beverage combined with 60 mg caffeine per 180 ml total beverage. The alcohol and caffeine will be mixed in a fruit punch beverage. Participants may self-administer as much beverage as they like with several constraints to assure safety (e.g., participants must stop drinking if their blood alcohol content is above .12 g/dl).
  Other Names: Alcohol 190 proof USP; Caffeine anhydrous USP
Drug: Alcohol + Caffeine-placebo — 14 g alcohol per 180 ml total beverage combined with 2.2 mg quinine per 180 ml total beverage. The alcohol and quinine will be mixed in a fruit punch beverage. Participants may self-administer as much beverage as they like with several constraints to assure safety (e.g., participants must stop drinking if their blood alcohol content is above .12 g/dl).
  Other Names: Alcohol 190 proof USP; Quinine hydrochloride dihydrate

SUMMARY:
The purpose of this study is to investigate the effects of caffeine on the self-administration of alcohol. The study will also examine the combined effects of alcohol and caffeine on behavioral performance, participant ratings of behavioral performance, and self-reported subjective effects.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of caffeine on alcohol self-administration. Volunteers will participate in 7 experimental sessions in which they will be given the opportunity to self-administer an alcohol + caffeine or alcohol + caffeine-placebo beverage. The first 6 sessions will involve exposure to the two beverage conditions in mixed order three times each (e.g., A, B, B, A, A, B). The seventh session will be a choice session in which the participant will make a single choice at the beginning of the session about which beverage they will consume that day. In addition to the primary outcomes of quantity of alcohol self-administered and beverage choice, three additional outcomes will be measured including: 1). indirect measures of reinforcing effects (e.g. subjective ratings of liking, well-being, take again); 2). an alcohol-sensitive behavioral measure; and 3). participant ratings of degree of behavioral impairment.

ELIGIBILITY:
Inclusion Criteria:

* Very light or moderate consumer of caffeine (either daily or non-daily).
* Social drinker of alcohol.
* Has experience in lifetime of heavy alcohol consumption.
* Read, write, and speak English fluently.

Exclusion Criteria:

* Serious and unstable illnesses including current hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, uncontrolled hypertension, and congestive heart failure), endocrinologic, neurologic (including stroke, transient ischemic attack, subarachnoidal bleeding, brain tumor, encephalopathy, and meningitis), or hematologic disease.
* Parkinson's disease, seizure disorder, or history of significant head trauma.
* Current psychiatric illness
* Pregnant or nursing women or women who are not using an effective means of birth control.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Total beverage consumed | Measured during 2.5 hour drinking period
  The primary outcome measure is the total volume of beverage consumed during alcohol + caffeine sessions and alcohol + caffeine-placebo sessions.

SECONDARY OUTCOMES:
Circular Lights Task | Approximately every 30 minutes of the 5.5 hour study period
  The Circular Lights Task is a measure of behavioral performance
The Biphasic Alcohol Effects Scale | Approximately every 30 minutes of the 5.5 hour study period
  The Biphasic Alcohol Effects Scale (BAES: Martin et al., 1993) will be repeatedly administered to assess changes in subjective alcohol effects over time. This measure is a commonly used 14-item scale that assesses stimulant (7 items) and sedative (7 items) subjective effects of drugs on a 10-point likert scale
Expired air breath alcohol measures | Approximately every 30 minutes during the 5.5 hour study period
  Breath alcohol measures will be taken repeatedly in order to assess blood alcohol levels, as well as assure safe discharge. In order to prevent mouth alcohol contamination of breath alcohol measurements, participants will be required to abstain from drinking for 5 minutes before each measurement and to rinse their mouth out thoroughly with water immediately before breath alcohol measures.
Subjective ratings 9-point likert scale | Approximately every 30 minutes during the 5.5 hour study period
  The following three questions will be asked on a 9-point likert scale:
  1. How much do you like the beverage you have been drinking today?
  2. Rate your sense of "well-being" right now.
  3. How much money would you be willing to pay for a standard mixed drink serving (e.g., 8 oz.) of this beverage at a bar?
Subjective ratings visual analogue scale | Approximately every 30 minutes during the 5.5 hour study period
  The following two questions will be answered on a visual analogue scale:
  1. How much do you want another drinking right now?
  2. How intoxicated do you feel?

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States